CLINICAL TRIAL: NCT03112408
Title: Coupling Between Adaptation of Saccadic Eye Movements and Visuo-spatial Perception and Attention Processes: a Behavioural Study in Humans.
Brief Title: Eye Movements and Visuo-spatial Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 69HCL17_0109; 2017-A00942-51 (Other: ID-RCB)
Record Dates: First submitted 2017-03-29; First posted 2017-04-13 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Cerebellum Disease
Keywords: cerebellar lesion; saccadic adaptation; spatial localization; visuo spatial perception; eye movements
MeSH Terms: conditions — Cerebellar Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- FORWARD (Axe 1) (Experimental)
  Interventions: Behavioral: Forward adaptation of reactive saccades
- BACKWARD (Axe 1) (Experimental)
  Interventions: Behavioral: Backward adaptation of reactive saccades
- CONTROL (Axe 1) (Experimental)
  Interventions: Behavioral: Execution of reactive saccades
- ADAPTATION (Axe 2) (Experimental)
  Interventions: Behavioral: Backward adaptation of reactive saccades
- CONTROL (Axe 2) (Experimental)
  Interventions: Behavioral: Generation of reactive saccades

INTERVENTIONS:
Behavioral: Forward adaptation of reactive saccades — Protocol of reactive saccade where the target is displaced in the same direction as the saccade in order to induce an adaptive increase of saccade amplitude ('forward adaptation')
  Arms: FORWARD (Axe 1)
Behavioral: Backward adaptation of reactive saccades — Protocol of reactive saccade where the target is displaced in a direction opposite to the saccade in order to induce an adaptive decrease of saccade amplitude ('backward adaptation')
  Arms: ADAPTATION (Axe 2); BACKWARD (Axe 1)
Behavioral: Execution of reactive saccades — Control protocol of reactive saccade with no displacement of the saccadic target (controlling for non specific factors possibly involved in forward and backward adaptation conditions)
  Arms: CONTROL (Axe 1)
Behavioral: Generation of reactive saccades — Control protocol of reactive saccade with no displacement of the saccadic target (controlling for non specific factors possibly involved in adaptation condition)
  Arms: CONTROL (Axe 2)

SUMMARY:
This research aims to highlight the key roles of the cerebellar and cortical fronto-parietal networks in the coupling of eye movements with visual perception and visuo-spatial attention.

DETAILED DESCRIPTION:
The first axe of this research focuses on the role of the cerebellum which has a major contribution to sensorimotor adaptation and more precisely in saccadic adaptation but the nature of this contribution is still debated. A classical assumption stipulates cerebellum has an exclusive action on saccadic burst generator in the brainstem whereas recent data increasingly support the view that cerebellum could also modulates cerebral cortex through a cerebello-thalamo-cortical pathway. On the other hand, several studies have shown that modification of saccade amplitude by saccadic adaptation leads to a distortion of the visual localization of briefly flashed spatial probes but no study to date has tested, the contribution of the cerebellum in these adaptation-induced mislocalizations. The main objective of this axe is to define the role of the cerebellum not only in saccadic adaptation, but also in mislocalizations which occur after adaptation. Moreover, in testing this assumption, arguments in favour -or in disfavor- of the action of the cerebellum on cortical stages dedicated to visuo-spatial perceptual processing will be provided. Besides, variability of cerebellar lesion (or cerebellar dysfunction) location in patients can lead to different pattern in saccadic adaptation and localization task performances. Identification of dissociations between these two abilities in some patients will define more precisely the role of the cerebellum in the coupling between saccadic adaptation and visuo spatial perception as an oculomotor plasticity territory and / or as a territory underlying the error signal coding generating this type of plasticity.

This second axe of this research aims to apply basic findings in healthy subject on the coupling between oculomotor plasticity and spatial attention to patients with parietal lesion, in order to evaluate a rehabilitation procedure for neglect patients. Habchi and colleagues showed that the adaptation of reactive saccades in the left hemifield has a boosting effect on attentional performance in the same hemifield. The coupling between these two mechanisms highlighted in healthy subjects can be used as fundamentals in the elaboration of a rehabilitation procedure for attentional disorders in the neglect syndrome. This syndrome is mainly observed after cerebral lesions in the right hemisphere, and is characterized by very disabling cognitive disorders such as an alteration of the spatial representation of left hemi-space and/or left hemi-body. stimulation of sensorimotor plasticity thanks to prismatic adaptation could be used as a rehabilitation procedure for this syndrome. Being another efficient way to stimulate sensorimotor plasticity, the equip believe that saccadic adaptation can also be used as a rehabilitation procedure for neglect patients. Moreover, due to its tight coupling with visual attention, the benefits of saccadic adaptation could be even stronger and longer lasting than the visuo-manual plasticity induced by prismatic adaptation.

ELIGIBILITY:
Inclusion Criteria:

* Age : from 18 to 80 ans included
* Visual acuity monocularly at distance and near corrected : > 5/10
* Possible understanding of experimental guidelines
* Possible respect for sustained seated position
* Subject covered by social security
* Agreement of the subject

Inclusion Criteria, specific to Axe 1:

* Cerebellar patients - Cerebellar degenerative disease (group A) or stroke (group B, délai depuis l'AVC : delay from the stroke : at least 1 month)

  * Scanner or MRI showing diffuse atrophy (group A) or focal cerebellar lesion (group B)
* Healthy subjects

  * Absence of known ophtalmological or neurological pathology

Inclusion Criteria, specific to Axe 2:

* Stroke patients - ischemic or hemorrhagic stroke

  * Encephalic MRI or CT scan showing an unique lesion
  * Minimal delay of one year after the stroke

Exclusion Criteria:

* Visual acuity monocularly < 5/10
* Language disorder restricting oral and reading comprehension of the study
* Severe disability limiting the maintenance of sitting position and concentration capacities for a period of 30 minutes consecutive
* Poor French language skills
* Non-stabilized medical condition
* Psychotropic medication intake
* Pregnant and / or nursing women
* Subject under guardianship or curatorship
* Subject frequently in healthcare or social care for purposes other than research
* Subject deprived of liberty by a judicial or administrative decision

Exclusion Criteria, specific to Axe 1:

• Cerebellar patients

- Disorders prohibiting the correct performance of the task (tremor, ocular instability)

Exclusion Criteria, specific to Axe 2:

• Stroke patients

* Hemianopsia homonima lateral
* Neurological degenerative disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Saccadic adaptation efficiency | At time of each experimental session, up to 2 months, since first experimental visit until last visit
  〖Adaptation〗_rate= (〖Amplitude 〗_post-〖Amplitude 〗_pre)/〖Amplitude 〗_pre

SECONDARY OUTCOMES:
Evolution of localization-task performances | At time of each experimental session, up to 2 months, since first experimental visit until last visit
  〖Improvement〗_performances= (〖Mislocalization 〗_post-〖Mislocalization 〗_pre)/〖Mislocalization 〗_pre
Evolution of attentional performances assessed by neuropsychological tests of neglect | At time of each experimental session, up to 2 months, since first experimental visit until last visit
  〖Improvement〗_performances= (〖Score 〗_post-〖Score〗_pre)/〖Score〗_pre

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Tilikete, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheviet A, Masselink J, Koun E, Salemme R, Lappe M, Froment-Tilikete C, Pelisson D. Cerebellar signals drive motor adjustments and visual perceptual changes during forward and backward adaptation of reactive saccades. Cereb Cortex. 2022 Sep 4;32(18):3896-3916. doi: 10.1093/cercor/bhab455. PMID 34979550